CLINICAL TRIAL: NCT07140263
Title: CARE-MI: A Comprehensive Group Intervention for Psychosocial Personnel at Risk of Experiencing Symptoms of Post-traumatic Stress and/or Moral Injury Associated With Work-related Stress: Design, Implementation, and Efficacy
Brief Title: A Comprehensive Group Intervention for Psychosocial Personnel at Risk of Stress and Moral Injury
Acronym: CARE-MI-PsychS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARE-MI-psychosocial personnel
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Moral Injury; TEPT
Keywords: psychosocial personnel; moral injury intervention; CARE-MI
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a multilevel randomized trial, in which preexisting work teams (group levels) are randomly assigned to either the CARE-MI intervention or a waitlist control group. Assessments are conducted at baseline, post-intervention, and at the 6-month follow-up.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARE MI (Experimental): CARE-MI is a trauma-informed integrative group intervention designed to reduce post-traumatic stress symptoms and moral injury in psychosocial personnel working with individuals with physical or mental health conditions.
  Interventions: Behavioral: CARE MI
- Waiting list (Delayed CARE-MI) (Other): Participants assigned to the waiting list will receive the CARE-MI intervention after the experimental group completes the initial study period. During the waiting period, they will receive usual institutional support. This design allows for comparison between groups while ensuring that all participants eventually receive the CARE-MI program.
  Interventions: Behavioral: CARE MI; Behavioral: TAU: Treatment as usual

INTERVENTIONS:
Behavioral: CARE MI — The intervention consists of four sessions, each lasting between 60 and 90 minutes, ideally delivered on consecutive weeks. It integrates psychoeducation on trauma and moral injury, emotional regulation strategies, and incorporates elements from several evidence-based approaches. These include the EMDR-IGTP-OTS group protocol, acceptance and values-based work from ACT, and self-compassion-focused interventions.
  In the Waiting List arm, CARE-MI will be delivered after the initial assessment period of the Experimental arm.
Behavioral: TAU: Treatment as usual — During the waiting period, Waiting list group will receive usual institutional support.
  Arms: Waiting list (Delayed CARE-MI)

SUMMARY:
The objective of this randomized controlled trial is to evaluate the effectiveness of the CARE-MI group intervention in reducing symptoms of post-traumatic stress and moral injury in support staff working with individuals diagnosed with physical or mental health conditions (psychosocial personnel). The study also seeks to assess its impact on symptoms of anxiety and depression, as well as its potential to improve overall well-being.

We will conduct a multicomponent study involving several pre-existing teams from collaborating centers, allowing the intervention to be evaluated in different institutional settings. This is a multilevel randomized trial, with each group randomly assigned, through blinded allocation using a computer program, to either the intervention group or a wait-list control group. Participants will be assessed at three time points: pre-intervention, post-intervention, and at a 6-month.

This trial is part of a larger research project that includes several related studies. Each study addresses a specific population and/or intervention, but all share the overarching aim of Coping and adaptation for recovery from moral injury.

DETAILED DESCRIPTION:
There is growing evidence of high prevalence rates of emotional distress, including PTSD, anxiety, depression, and moral injury, among healthcare professionals, particularly those exposed to high emotional loads or critical care settings. Studies report PTSD rates ranging from 10% to 20%, and up to 30% in ICU staff. These figures increase significantly during large-scale crises such as pandemics. For instance, during the COVID-19 outbreak, rates of PTSD symptoms reached up to 54% among U.S. healthcare workers, along with 48% for depression and 30% for anxiety. Similar findings were observed in Spain and China, with high moral injury prevalence associated with anxiety and depression symptoms.

Moral injury is particularly concerning in settings with staffing shortages, where professionals feel unable to provide adequate care. This scenario extends to the mental health support network, including social and psychological care teams. In Spain, significant rates of emotional exposure (36%) and workplace violence have been reported among technical and support staff.

Although trauma-focused interventions have shown efficacy in treating PTSD, most evidence focuses on individual formats. Group interventions, however, offer a scalable, resource-efficient alternative, with promising outcomes reported for ACT, mindfulness, EMDR, and other trauma-informed approaches.

Despite this evidence, few interventions are specifically adapted and evaluated for mental health and healthcare professionals in their specific work contexts. This trial addresses this gap by evaluating the CARE-MI protocol in real-world care settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Be currently employed as healthcare or support staff at the time of the intervention
* Provide informed consent
* Be fluent in Spanish

Exclusion Criteria:

- None explicitly defined

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in posttraumatic stress symptoms | Time Frame: Baseline, post-intervention (4 weeks), 6-month follow-up
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5; Blevins et al., 2015). Higher scores indicate greater PTSD symptoms (minimum and maximun values: 0 and 80).
Change in moral injury symptoms | [Time Frame: Baseline, post-intervention (4 weeks), 6-month follow-up]
  Healthcare Moral Injury Scale (HMIS; Fradley et al., under review). Higher scores indicate higher levels of moral injury (minimum and maximun values: 5 and 50).

SECONDARY OUTCOMES:
Change in anxiety symptoms | [Time Frame: Baseline, post-intervention (4 weeks), 6-month follow-up]
  Generalized Anxiety Disorder 7-item scale (GAD-7; Spitzer et al., 2006). Higher scores indicate greater anxiety (minimum and maximun values: 0 and 21).
Change in depressive symptoms | [Time Frame: Baseline, post-intervention (4 weeks), 6-month follow-up]
  Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001). Higher scores indicate greater depressive symptoms (minimum and maximun values: 0 and 27).
Change in mental wellbeing | [Time Frame: Baseline, post-intervention (4 weeks), 6-month follow-up]
  Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS; Tennant et al., 2007). Higher scores indicate better wellbeing (minimum and maximun values: 14 and 70)..
Change in perceived meaning at work | Time Frame: Baseline
  Work and Meaning Inventory (WAMI; Steger, 2012). Higher scores indicate greater perceived meaning (minimum and maximun values: 10 and 50).
Change in perceived ability to cope with trauma | [Time Frame: Baseline, post-intervention (4 weeks), 6-month follow-up]
  Perceived Ability to Cope with Trauma Scale (PACT; Bonanno et al., 2011). Higher scores indicate greater coping flexibility (minimum and maximun values: 20 and 140).
Change in openness to the future | [Time Frame: Baseline, post-intervention (4 weeks), 6-month follow-up]
  Openness to the Future Scale (OFS; Botella et al., 2018). Higher scores indicate greater positive affective orientation toward the future (minimum and maximun values: 10 and 50).
Change in experiential avoidance | [Time Frame: Baseline, post-intervention (4 weeks), 6-month follow-up]
  Brief Experiential Avoidance Questionnaire (BEAQ; Gámez et al., 2014). Higher scores indicate greater experiential avoidance (minimum and maximun values: 15 and 90).
Satisfaction with the intervention | [Time Frame: Post-intervention (4 weeks)]
  Client Satisfaction Questionnaire-8 (CSQ-8; Larsen et al., 1979). Higher scores indicate greater satisfaction with the intervention (minimum and maximun values: 4 and 32).

CONTACTS AND LOCATIONS:
Overall Officials: Regina Espinosa, Full Porfessor, Principal Investigator — Camilo Jose Cela University; Carmen Valiente, Full Porfessor, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code